CLINICAL TRIAL: NCT05488483
Title: A Feasibility Study of Multispectral Optoacoustic Tomography (MSOT) Imaging in Patients With Tumors
Brief Title: A Study of Tumor Imaging With Multispectral Optoacoustic Tomography
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-374
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Melanoma
Keywords: Multispectral Optoacoustic Tomography Imaging; MSOT; Memorial Sloan Kettering Cancer Center; 21-374
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast and Melanoma Cohort: Participants with a suspicious finding at breast ultrasonography (BI-RADS 4 suspicious abnormality; BI-RADS 5, highly suggestive for malignancy) who are scheduled for ultrasound-guided breast biopsy will undergo MSOT imaging of the suspicious breast tumor detected with ultrasound imaging and any additional lesion present in either breast before undergoing ultrasound-guided breast biopsy as the standard of care. We will evaluate MSOT in 10 patients from the Melanoma Surgical Oncology Clinics (Dr. Ariyan, Co-I) with pathologically confirmed ITM following physical exam and biopsy. We will also evaluate MSOT in five melanoma patients with pathologically confirmed IT metastases scheduled for neoadjuvant immunotherapy prior to surgical resection.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography Imaging

INTERVENTIONS:
Diagnostic Test: Multispectral Optoacoustic Tomography Imaging — Each participants will undergo MSOT imaging of the suspicious breast tumor detected with ultrasound imaging and any additional lesion present in either breast before undergoing ultrasound-guided breast biopsy as the standard of care. Melanoma participants with pathologically confirmed ITM will undergo MSOT imaging following physical exam and biopsy. Melanoma patients receiving immunotherapy will undergo MSOT imaging prior to and following immunotherapy.
  Other Names: MSOT

SUMMARY:
Participants in this study will have Multispectral Optoacoustic Tomography/MSOT imaging of both breasts immediately before their ultrasound-guided breast biopsy procedure begins. After the MSO imaging is completed, participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a female or male who is 18 years of age or older.
* Participant must meet one of the following:

  * Suspicious breast imaging finding detected on either mammography, ultrasound, or MRI that is visible on ultrasound and therefore recommended for ultrasound-guided breast biopsy (BI-RADS 4 suspicious abnormality; BI-RADS 5, highly suggestive for malignancy)
  * No previous treatment for breast cancer
  * Diagnosis of melanoma

Exclusion Criteria:

* Life expectancy < 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a suspicious breast imaging finding detected on either mammography, ultrasound or MRI that is visible on ultrasound and therefore recommended for ultrasound-guided breast biopsy (BI-RADS 4 suspicious abnormality; BI-RADS 5, highly suggestive for malignancy) who are scheduled for ultrasound-guided breast biopsy by the Memorial Sloan Kettering Department of Radiology Breast Imaging Service will be included.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants where tumors were visualized | 1 year
  The primary goal of this study is to evaluate the feasibility of MSOT for breast cancer and melanoma detection. Feasibility is defined as the ability of the method to visualize tumors that have been identified with standard methods (ultrasound, mammography, MRI), and the ability to obtain oxygenation maps of benign and malignant breast and melanoma tumors. MSOT will be considered feasible if it is able to visualize tumors and obtain oxygenation maps in at least 14 patients out of 20

CONTACTS AND LOCATIONS:
Overall Officials: Jan Grimm, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (3):
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
- Helmholtz Institute (Data Analysis Only), Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org